CLINICAL TRIAL: NCT00307593
Title: Infliximab Versus Rituximab in Systemic Necrotizing Vasculitides With Positive ANCA After Relapse or Resistant Immunosuppressant Therapies
Brief Title: RATTRAP: Infliximab Versus Rituximab in Systemic Necrotizing Vasculitides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P020931; AOM02098
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-03

CONDITIONS: Wegener's Granulomatosis; Churg-Strauss Syndrome; Microscopic Polyangiitis
Keywords: Systemic ANCA+ vascularizes; Relapse; Corticosteroids; Immunosuppressant; Infliximab/rituximab; Patients with relapsing or refractory forms of ANCA; associated vasculitides Microscopic polyangiitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Churg-Strauss Syndrome; Microscopic Polyangiitis; Recurrence | interventions — Infliximab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Rituximab
  Interventions: Drug: Rituximab
- 2 (Active Comparator): Infliximab
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab
  Arms: 2
Drug: Rituximab — Rituximab
  Arms: 1

SUMMARY:
The purpose of this study is to compare a 2 immunosuppressant regimen for the treatment of relapsing or refractory necrotizing antineutrophil cytoplasmic antibody (ANCA) associated vasculitides.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of rituximab versus infliximab in relapsing or refractory forms of ANCA+ vasculitides (Microscopic Polyangiitis, Wegener's granulomatosis and Churg-Strauss syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Systemic ANCA positive (+) vasculitides
* Relapsing or refractory vasculitides, resistant to corticosteroids and reference immunosuppressant therapies
* Age >18 years old
* Written informed consent

Exclusion Criteria:

* Newly diagnosed patient
* Patient that had never received an immunosuppressant before to treat his/her vasculitis
* Malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Partial or complete remission of the vasculitides | one year

SECONDARY OUTCOMES:
To study the safety and adverse effects of both regimens | one year
Microscopic polyangiitis | one year
Wegener's granulomatosis | one year
Churg-Strauss syndrome | one year

CONTACTS AND LOCATIONS:
Overall Officials: Loïc GUILLEVIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France